CLINICAL TRIAL: NCT02089867
Title: A Randomized Open Label Trial to Assess the Effect of Plant Sterols Associated With Ezetimibe in LDL-cholesterol Levels in Coronary Patients Previously on Statin Therapy
Brief Title: Plant Sterols Effect on Previous Statin Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jose Rocha Faria Neto (Other)
Responsible Party: Sponsor-Investigator, Jose Rocha Faria Neto, Professor in Medicine, Pontifícia Universidade Católica do Paraná (PUCPR), Pontifícia Universidade Católica do Paraná
Organization: Pontifícia Universidade Católica do Paraná (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 632
Record Dates: First submitted 2014-03-15; First posted 2014-03-18 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: Ezetimibe; Plant sterol; Hydroxymethylglutaryl coenzyme A Reductase Inhibitors; Coronary artery disease; LDL-cholesterol
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ezetimibe; Phytosterols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ezetimibe (Experimental): The ezetimibe group will receive 10 mg/day ezetimibe for 6 weeks.
  Interventions: Drug: Ezetimibe
- Plant sterols (Experimental): The plant sterol group will receive spread enriched with 2g daily of plant sterols for 6 weeks
  Interventions: Dietary Supplement: Plant sterols
- Control group (No Intervention): No additional therapy, statin maintenance
- Ezetimibe + plant sterols (Experimental): The ezetimibe + plant sterols group will receive ezetimibe 10 mg/day + spread enriched with 2g daily of plant sterols for 6 weeks
  Interventions: Other: Ezetimibe + plant sterols

INTERVENTIONS:
Other: Ezetimibe + plant sterols — The ezetimibe + plant sterols group will receive ezetimibe 10 mg/day + spread enriched with 2g daily of plant sterols for 6 weeks
  Arms: Ezetimibe + plant sterols
Drug: Ezetimibe — The ezetimibe group will receive 10 mg/day ezetimibe for 6 weeks.
  Arms: Ezetimibe
Dietary Supplement: Plant sterols — The plant sterol group will receive spread enriched with 2g daily of plant sterols for 6 weeks
  Arms: Plant sterols

SUMMARY:
The purpose of this study is to determine the effect of plant sterols associated with ezetimibe in LDL-cholesterol levels in coronary patients previously on statin therapy

DETAILED DESCRIPTION:
Background: Consumption of food products enriched with plant sterols and treatment with ezetimibe both reduce cholesterol absorption in the intestine by different mechanisms and effectively reduce LDL cholesterol (LDL-c) plasma levels. Although, the associated usage of ezetimibe to plants sterols in coronary patients not reaching recommended lipid levels despite the use of statins has not yet been demonstrated. Objectives: Evaluate if ezetimibe 10mg associated to plant sterols spread enriched with 2g of plant sterols in coronary patients not reaching recommended lipid levels despite the use of statins is able to reduce cholesterol levels after 6 week treatment. Methods: Prospective, open-label study with both male and female patients with stable coronary disease and LDL > 70mg/dL. Patients will be randomized for the following 6 week treatment: control group (CT) no additional statin therapy, ezetimibe group (EZ) 10 mg/day ezetimibe, plant sterol group (PS) spread enriched with 2g of plant sterols or ezetimibe+plant sterols group (EZ+PS) 10mg/day EZ + 2g PS. Anthropometric evaluations and laboratory exams (blood glucose test, total cholesterol, LDL-c, HDL-c, triglycerides, and C-Reactive Protein) will be performed in all groups at baseline and after the sixth week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous myocardial infarction, stroke or coronary angiography demonstrating significant coronary disease.
* Subjects under statin treatment with a fixed dosage for the previous three months before randomization, and did not reached LDL less than 70mg/dl.

Exclusion Criteria:

* Subjects already taking ezetimibe and/or plant sterols
* Younger than 18 years
* Presence of any contraindication to statin
* Pregnant women or breast-feeding women or
* Patients with previous history of statin hypersensibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Decrease of LDL cholesterol levels due to plant sterols associated with ezetimibe. | 6 weeks
  The primary end-point was the LDL cholesterol levels change after the plant sterols associated with ezetimibe from baseline up to 6 week treatment.

SECONDARY OUTCOMES:
Any change of non-LDL-cholesterol, total cholesterol, high-density lipoprotein (HDL), very-low-density lipoprotein (VLDL), triglycerides levels, and changes in high sensitive C reactive protein (CRP) levels. | 6 weeks
  Secondary end points included any change of non-LDL-cholesterol, total cholesterol, high-density lipoprotein (HDL), very-low-density lipoprotein (VLDL), triglycerides levels, and changes in high sensitive C reactive protein (CRP) levels from baseline up to 6 week treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Faria Neto, PhD, Study Chair — Professor in Medicine, Pontifícia Universidade Católica do Paraná (PUCPR)
Locations (1):
- Jose Rocha Faria Neto, Curitiba, Paraná, Brazil